CLINICAL TRIAL: NCT02743819
Title: Phase II Study of Pembrolizumab and Ipilimumab Following Initial Anti-PD1/L1 Antibody
Brief Title: Pembrolizumab and Ipilimumab After Prior Immunotherapy for Melanoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB17-0686; IRB15-1788 (Other: University of Chicago)
Record Dates: First submitted 2016-04-14; First posted 2016-04-19 (Estimated); Results first posted 2022-04-21 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Melanoma
Keywords: Melanoma; Pembrolizumab; Ipilimumab
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab; Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Treatment with the combination of pembrolizumab and ipilimumab.
  Interventions: Drug: Pembrolizumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab given every 3 weeks (200 mg) by IV infusion.
  Other Names: Keytruda
Drug: Ipilimumab — Ipilimumab given every 3 weeks (200 mg) by IV infusion for total of 4 doses.
  Other Names: Yervoy

SUMMARY:
Phase II study evaluating the benefit of the combination of anti-PD1 (pembrolizumab) and anti-CTLA4 (ipilimumab) antibodies in advanced melanoma. The study will determine the response rate of the combination and evaluate other clinical parameters such as progression-free survival and safety of the combination following anti-PD1/L1 antibody. The study will also provide the opportunity to investigate blood or tumor based factors that may predict response to anti-PD1 antibody in combination with anti-CTLA4.

DETAILED DESCRIPTION:
Primary Objective:

To determine the irRECIST* response rate of pembrolizumab with ipilimumab following initial progression or stable disease to anti-PD1/L1 antibody (or combination not containing anti-CTLA4) in subjects with advanced melanoma.

Secondary Objective

1. To summarize the progression-free survival (RECIST v1.1 and irRC) of the combination following prior treatment with anti-PD1/L1 antibody.
2. To assess the safety of the combination following prior treatment with anti-PD1/L1 antibody.

Exploratory Objective:

To evaluate changes in the tumor microenvironment and other biospecimens before and after adding ipilimumab to pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible for participation in this trial, the subject must:

1. Be willing and able to provide written informed consent for the trial.
2. Be 18 years of age on day of signing informed consent.
3. Have experienced disease progression or stable disease lasting at least 24 weeks during treatment with an anti-PD1/L1 antibody as the treatment regimen immediately prior to accrual to this study or disease progression within 6 months of adjuvant anti-PD1 antibody.
4. Have measurable disease based on irRECIST 1.1.
5. Have a performance status of 0 or 1 on the ECOG Performance Scale.
6. Demonstrate adequate organ function as defined below, all screening labs should be performed within 10 days of treatment initiation.

   Hematological Absolute neutrophil count (ANC) ≥1,500 /mcL Platelets ≥100,000 / mcL Hemoglobin ≥8 g/dL or ≥4.96 mmol/L

   Renal Serum creatinine OR Measured or calculated creatinine clearance ≤1.5 X upper limit of normal (ULN) OR ≥60 mL/min for subject with creatinine levels > 1.5 X institutional ULN (GFR can also be used in place of creatinine or CrCl)

   Hepatic Serum total bilirubin ≤ 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR ≤ 5 X ULN for subjects with liver metastases Albumin >2.5 mg/dL

   Coagulation International Normalized Ratio (INR) or Prothrombin Time (PT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

   Activated Partial Thromboplastin Time (aPTT) ≤1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
7. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
8. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
9. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Exclusion Criteria:

The subject must be excluded from participating in the trial if the subject:

1. Has received study therapy (including investigational device) as part of a clinical trial within 4 weeks of the first dose of treatment, with the exclusion of an anti-PD1/L1 antibody given as either a single agent or non-CTLA-4 antibody containing combination.
2. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
3. Has a known history of active TB (Bacillus Tuberculosis)
4. Hypersensitivity to pembrolizumab or any of its excipients.
5. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 (excluding commercial or investigational anti-PD1 or anti-PD-L1 antibodies as single agents) or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
6. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
7. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
8. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
9. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
10. Patients with uveal/ocular melanoma are excluded.
11. Has known history of, or any evidence of active, non-infectious pneumonitis.
12. Has an active infection requiring systemic therapy.
13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
15. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
16. Has received prior therapy with an anti-CTLA4 agent.
17. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
18. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
19. Has received a live vaccine within 30 days of planned start of study therapy.

Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines are live attenuated vaccines, and are not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-06-28 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2026-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Gajewski, M.D., Principal Investigator — University of Chicago
Locations (10):
- United States (10):
  - University of South Alabama, Mobile, Alabama
  - Mount Sinai Medical Center of Florida, Miami Beach, Florida
  - H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida
  - University of Chicago, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - NorthShore University HealthSystem, Evanston, Illinois
  - Oncology Specialists S.C., Park Ridge, Illinois
  - Illinois Cancer Care, Peoria, Illinois
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - Virginia Commonwealth University/ Massey Cancer Center, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started (70 patients enrolled in the study and received at least one dose of study treatment.) | 70
Completed | 62
Not Completed | 8
Not completed — Lack of Efficacy | 5
Not completed — Death | 2
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment
Number analyzed (Participants) | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 36
Age, Continuous [Median (Full Range); unit: years] | 64 [27 to 87]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 47
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 68
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 68
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 70

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (OR) Per irRECIST
Description: Per Response Evaluation Criteria for use in trials testing immunotherapeutics (iRECIST) for target lesions and assessed by CT or MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 70
Participants | 20

2. Secondary Outcome: Progression Free Survival Using the Kaplan Meier Method
Description: Time to disease progression or death. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: 24 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment
Number analyzed (Participants) | 70
months | 5 [2.8 to 8.3]

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Any treatment-related adverse event
Time Frame: 30 days after the end of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 70
Participants | 62

ADVERSE EVENTS:
Time Frame: Adverse event data was followed for each patient from receiving their first dose of study therapy up through two years following drug discontinuation.
Description: Adverse events were reported according to Common Terminology Criteria for Adverse Events (CTCAE) version 4.0.
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 28/70
Serious Adverse Events (participants affected / at risk) | 20/70
Other Adverse Events (participants affected / at risk) | 62/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=70)
Abdominal pain (Gastrointestinal disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 1
Bone infection (Infections and infestations) | 1
Colitis (Gastrointestinal disorders) | 2
Colonic perforation (Gastrointestinal disorders) | 1
Confusion (Psychiatric disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Esophageal obstruction (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 2
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal disorders - other (Gastrointestinal disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Hematoma (Vascular disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 1
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Lung infection (Infections and infestations) | 1
Nausea (Gastrointestinal disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Sepsis (Infections and infestations) | 2
Skin and subcutaneous tissue disorders - other (Skin and subcutaneous tissue disorders) | 1
Skin infection (Infections and infestations) | 1
Stroke (Nervous system disorders) | 1
Surgical and medical procedures - other (Surgical and medical procedures) | 2
Thromboembolic event (Vascular disorders) | 1
Vestibular disorder (Ear and labyrinth disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (N=70)
Abdominal pain (Gastrointestinal disorders) | 13
Adrenal insufficiency (Endocrine disorders) | 5
Alanine aminotransferase increased (Investigations) | 14
Alkaline phosphatase increased (Investigations) | 8
Anemia (Blood and lymphatic system disorders) | 17
Anorexia (Metabolism and nutrition disorders) | 16
Arthralgia (Musculoskeletal and connective tissue disorders) | 11
Aspartate aminotransferase increased (Investigations) | 11
Back pain (Musculoskeletal and connective tissue disorders) | 8
Bloating (Gastrointestinal disorders) | 9
Bruising (Injury, poisoning and procedural complications) | 4
Chills (General disorders) | 4
Colitis (Gastrointestinal disorders) | 5
Constipation (Gastrointestinal disorders) | 19
Cough (Respiratory, thoracic and mediastinal disorders) | 13
Creatinine increased (Investigations) | 8
Dehydration (Metabolism and nutrition disorders) | 8
Diarrhea (Gastrointestinal disorders) | 34
Dizziness (Nervous system disorders) | 8
Dry mouth (Gastrointestinal disorders) | 7
Dysgeusia (Nervous system disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 16
Edema limbs (General disorders) | 8
Endocrine disorders - other (Endocrine disorders) | 4
Fatigue (General disorders) | 26
Fever (Gastrointestinal disorders) | 7
Flatulence (Gastrointestinal disorders) | 8
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 10
Headache (Nervous system disorders) | 16
Hot flashes (Vascular disorders) | 6
Hyperglycemia (Metabolism and nutrition disorders) | 5
Hyperkalemia (Metabolism and nutrition disorders) | 17
Hypertension (Vascular disorders) | 14
Hypoalbuminemia (Metabolism and nutrition disorders) | 13
Hypocalcemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 5
Hyponatremia (Metabolism and nutrition disorders) | 7
Hypothyroidism (Endocrine disorders) | 10
Hypotension (Vascular disorders) | 6
Infections and infestations - other (Infections and infestations) | 4
Insomnia (Psychiatric disorders) | 9
Investigations - other (Investigations) | 7
Lipase increased (Investigations) | 4
Lymphocyte count decreased (Investigations) | 17
Memory impairment (Nervous system disorders) | 4
Musculoskeletal and connective tissue disorder - other (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 9
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6
Nausea (Gastrointestinal disorders) | 23
Neoplasms benign, malignant and unspecified - other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5
Nervous system disorders - other (Nervous system disorders) | 4
Neuropathy-sensory (Nervous system disorders) | 7
Pain (General disorders) | 9
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4
Platelet count decreased (Investigations) | 6
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 4
Pruritis (Skin and subcutaneous tissue disorders) | 29
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 23
Serum amylase increased (Investigations) | 4
Sinus bradycardia (Cardiac disorders) | 7
Skin and subcutaneous tissue disorders - other (Skin and subcutaneous tissue disorders) | 5
Thromboembolic event (Vascular disorders) | 7
Upper respiratory infection (Infections and infestations) | 6
Urinary frequency (Renal and urinary disorders) | 5
Urinary tract infection (Infections and infestations) | 6
Vomiting (Gastrointestinal disorders) | 18
Weight gain (Investigations) | 5
Weight loss (Investigations) | 12
White blood cell decreased (Investigations) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-10): https://cdn.clinicaltrials.gov/large-docs/19/NCT02743819/Prot_SAP_000.pdf